CLINICAL TRIAL: NCT00272948
Title: Prospective Randomized Study of the Incidence and Outcome of Veno-Occlusive Disease (VOD) With the Prophylactic Use of Defibrotide (DF) in Pediatric Stem Cell Transplantation
Brief Title: Pediatric Trial Investigating the Incidence & Outcome of Veno-Occlusive Disease With the Prophylactic Use of Defibrotide
Acronym: VOD-DF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Jazz Pharmaceuticals (Industry); Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Liz Clark, European Group for Blood and Marrow Transplantation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EudraCT Number:2004-000592-33; EBMT-PD-200601
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Hepatic Veno-Occlusive Disease
Keywords: Venoocclusive disease; Pediatric; myeloablative conditioning; stem cell transplant
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease | interventions — defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylaxis Arm (Experimental)
  Interventions: Drug: Defibrotide
- Control Arm (Active Comparator)
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — Defibrotide 25 mg/kg/d
Drug: Defibrotide — Defibrotide 25 mg/kg/d iv in 4 doses beginning at day of conditioning until day +30 or until discharge from inpatient care (with a minimum treatment of 14 days) if VOD does not occur.
  Arms: Prophylaxis Arm
Drug: Defibrotide — Defibrotide 25 mg/kg/d iv therapeutically when patients fulfil modified Seattle criteria
  Arms: Control Arm

SUMMARY:
The aim of this trial is to evaluate whether the prophylactic use of Defibrotide (DF) in pediatric patients (age less than 18 years) undergoing stem cell transplantation and who are at high risk of developing hepatic Veno-occlusive Disease (VOD) will have an impact on the incidence and severity of the disease. Patients will be randomly assigned to one of two treatment arms: Those allocated to the Prophylactic Arm will receive the study drug (Defibrotide) from the day of conditioning onwards. Patients allocated to the Control Arm will receive the study drug (Defibrotide) from the day that VOD is diagnosed.

DETAILED DESCRIPTION:
Comparison/control intervention and duration of the intervention:

Patients will be assigned randomly to either the Defibrotide (DF) prophylaxis arm or the control arm. Those allocated to the DF prophylaxis arm (DF 25 mg/kg/d iv in 4 doses) will begin treatment at day of conditioning and stop at day +30 after Stem Cell Transplantation (SCT) or upon discharge from inpatient care. There is no dose adjustment for a patient of the study arm who developed VOD, they continue with the 25mg/kg/d iv.

Patients allocated to the control arm receive no prophylactic measures and will start DF (25 mg/kg/d iv in 4 doses) beginning at day of diagnosis of Veno-occlusive Disease (VOD) according to modified Seattle criteria. Treatment will be stopped at complete resolution of symptoms. In both arms patients who developed VOD will continue DF until:

* complete resolution of the ascites and
* reversion of the hepatopedal flow (if present) and
* normalization of the total and direct bilirubin

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years
* myeloablative conditioning and autologous or allogeneic stem cell transplantation with at least one of the following risk factors for VOD:

  1. Pre-existing liver disease
  2. Second myeloablative HSCT
  3. History of treatment with gemtuzumab ozogamicin (MYLOTARGÒ, GO, CMA-676, Wyeth)
  4. Allogeneic HSCT for leukemia beyond the second relapse
  5. Osteopetrosis (OP)
  6. Conditioning with busulfan and melphalan
  7. Macrophage activating syndromes (MAS, like hemophagocytic lymphohistiocytosis, Griscelli, Chediak-Higashi
  8. Adrenoleukodystrophy (ALD)

Exclusion Criteria:

* Pregnant patients
* Patients who are transplanted but do not fulfill any of the above mentioned criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2005-12; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate if prophylactic DF has an impact on the incidence of VOD | Day + 30 post HSCT

SECONDARY OUTCOMES:
Occurrence of Multi-System Organ Failure and Survival (all causes of mortality) | day +100 post HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Selim Corbacioglu, MD, Principal Investigator — University of Ulm, Germany
Locations (30):
- Austria (2):
  - University Hospital, Graz
  - St Anna Kinderspital, Vienna
- Inst. Gustave Roussy, Villejuif, France
- Germany (11):
  - University Hospital, Dresden
  - Klinik Kinder-Onkologie, Düsseldorf
  - Johann-Wolfgang Goethe Universität, Frankfurt
  - Universitätsspital Eppendorf, Hamburg
  - Medical School, Hanover
  - University Hospital, Heidelberg
  - Kinderklinik, Jena
  - Christian-Albrecht -University, Kiel
  - Kinderpoliklinik Uni, München
  - Poliklinik Kinderheilkunde, Münster
  - Universitätsspital, Tübingen
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- Schneider Children's MC, Petah Tikva, Israel
- Italy (3):
  - Institute G. Gaslini, Genova
  - Ospedale S. Gerardo, Monza
  - Clinica di Oncoematologia Pediatrica, Padua
- University Hospital, Utrecht, Netherlands
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - University Hospital, Huddinge
  - University Hospital, Lund
  - University Hospital, Uppsala
- Switzerland (4):
  - University Children Hospital, Basel
  - Inselspital, Bern
  - Hopital Cantonal Universitaire, Geneva
  - University Hospital, Zurich
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - Children's Hospital, Manchester

REFERENCES:
- [Derived] Corbacioglu S, Grupp SA, Richardson PG, Duarte R, Pagliuca A, Ruutu T, Mahadeo K, Carreras E. Prevention of veno-occlusive disease/sinusoidal obstruction syndrome: a never-ending story and no easy answer. Bone Marrow Transplant. 2023 Aug;58(8):839-841. doi: 10.1038/s41409-023-02007-2. Epub 2023 May 25. No abstract available. PMID 37231094
- [Derived] Corbacioglu S, Cesaro S, Faraci M, Valteau-Couanet D, Gruhn B, Rovelli A, Boelens JJ, Hewitt A, Schrum J, Schulz AS, Muller I, Stein J, Wynn R, Greil J, Sykora KW, Matthes-Martin S, Fuhrer M, O'Meara A, Toporski J, Sedlacek P, Schlegel PG, Ehlert K, Fasth A, Winiarski J, Arvidson J, Mauz-Korholz C, Ozsahin H, Schrauder A, Bader P, Massaro J, D'Agostino R, Hoyle M, Iacobelli M, Debatin KM, Peters C, Dini G. Defibrotide for prophylaxis of hepatic veno-occlusive disease in paediatric haemopoietic stem-cell transplantation: an open-label, phase 3, randomised controlled trial. Lancet. 2012 Apr 7;379(9823):1301-9. doi: 10.1016/S0140-6736(11)61938-7. Epub 2012 Feb 23. PMID 22364685
- See also: sponsor's Web site — http://www.ebmt.org